CLINICAL TRIAL: NCT00475722
Title: A Mediterranean Diet in Colon Cancer Prevention
Brief Title: Healthy Eating for Colon Cancer Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Zora Djuric, Research Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00007622
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2015-07-08 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-08

CONDITIONS: Colon Cancer
Keywords: cancer; colon; prevention; healthy eating; Mediterranean diet; PGE2; cyclooxygenase; lipoxygenase; Healthy People 2010 diet; dietary prevention of colon cancer
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Healthy Eating (Active Comparator): Healthy People 2010 Diet using an exchange list
  Interventions: Behavioral: 1 Healthy Eating
- 2 Mediterranean (Experimental): Mediterranean Diet using an exchange list
  Interventions: Behavioral: 2 Mediterranean

INTERVENTIONS:
Behavioral: 1 Healthy Eating — 6 months telephone counseling
  Arms: 1 Healthy Eating
Behavioral: 2 Mediterranean — 6 months telephone counseling
  Arms: 2 Mediterranean

SUMMARY:
The purpose of this study is to help develop diets for colon cancer prevention. This study will compare the Mediterranean diet to the Healthy People 2010 diet in 120 subjects with increased risk for colorectal cancer.

DETAILED DESCRIPTION:
There is substantial epidemiological evidence that dietary patterns influence colorectal cancer risk. The associations of any particular nutrient with increased or decreased risks, however, may not be due to that nutrient per se but to the whole foods that are rich in that nutrient. Simultaneously, reducing intakes of foods associated with increased risk while increasing foods identified in preventive diets may be the best approach for prevention. The Cretan-Mediterranean diet in particular appears to hold great promise for cancer prevention. The major components of the traditional Cretan diet have been associated with decreased colon cancer. Relative to the American diet, this diet has lower n-6/n-3 and n-6/n-9 fatty acid ratios, lower polyunsaturated fatty acid intake, lower red meat intake, and higher intakes of plant-based foods and monounsaturated fatty acids.

The hypothesis of this study is that adherence to a Mediterranean type of diet will result in a decrease in n-6 fatty acids and increased n-3 and n-9 fatty acids in human colorectal mucosa. This together with aspects of the diet such as increased intakes of fruits and vegetables, is expected to modulate eicosanoid metabolism and epithelial proliferation in normal mucosa. 120 persons, with an increased risk for colorectal cancer, will be randomized to a modified Mediterranean diet or a Healthy People 2010 diet for six months.

ELIGIBILITY:
Inclusion Criteria:

* Prior adenomatous polyp.
* Prior resected early (Dukes A, B, or C) colon cancer. With the exception of curative surgery for small lesions, such as endoscopically removed cancers, eligible subject will be at least two years post treatment for colorectal cancer.
* A history of colon cancer in a primary relative or in two secondary relatives.
* Good general health and not expecting major lifestyle changes in the next 6 months.
* Age 21 or older.
* Not expecting a change in hormonal therapies over the next 6 months.
* Taking less than 81 mg/day or 325 mg aspirin every other day for prevention of cardiovascular disease.
* Dietary intake that is within the usual range for a typical American diet.
* Read and understand English.
* Sign the consent and willing to comply with all study procedures.
* Have a telephone.
* At least 5 years post any type of treatment for any other cancer except cancers that were removed completely by surgery and no other treatment was undergone.
* No more than occasional use (< 25% of the time) of pain medications and willing to take only regular strength acetaminophen while on study except for 81 mg/day or 325 mg every other day of aspirin for prevention of cardiovascular disease.

Exclusion Criteria:

* On medically prescribed diets or following a diet that would require extensive counseling to correct nutritional deficiencies.
* Taking supplements or medications that might obscure our ability to detect an effect of diet (eg. lipid-lowering medications, insulin, fish oils, mega-vitamins).
* Are pregnant or lactating or planning to get pregnant.
* Previous diagnosis of HIV or hepatitis C.
* Have cancer at the present time.
* Being treated with or taking therapies or supplements that could obscure our ability to detect diet effects, such as fish oils.
* Previous advanced cancer (Duke's D) or hereditary and familial polyposis (HNPCC/FAP) because the latter are rare conditions with unique etiology.
* Due to the effects of inflammation on biomarker levels in mucosa, persons with Crohn's disease or inflammatory bowel disease will be excluded.
* Persons with BMI < 18.5 or > 35 kg/m2 since low BMI could indicate eating disorders and high BMI values, above the midpoint of the obesity range, could indicate more prevalent health problems and these persons can be more difficult to counsel.
* Persons taking very high levels of aspirin or non-steroidal anti-inflammatory agents (NSAIDS) for conditions such as arthritis, a chronic inflammatory condition, will be excluded since it will preclude our ability to detect a further decrease in PGE2.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zora Djuric, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Djuric Z, Ruffin MT 4th, Rapai ME, Cornellier ML, Ren J, Ferreri TG, Askew LM, Sen A, Brenner DE, Turgeon DK. A Mediterranean dietary intervention in persons at high risk of colon cancer: recruitment and retention to an intensive study requiring biopsies. Contemp Clin Trials. 2012 Sep;33(5):881-8. doi: 10.1016/j.cct.2012.05.006. Epub 2012 May 26. PMID 22640923
- [Result] Sidahmed E, Cornellier ML, Ren J, Askew LM, Li Y, Talaat N, Rapai MS, Ruffin MT, Turgeon DK, Brenner D, Sen A, Djuric Z. Development of exchange lists for Mediterranean and Healthy Eating diets: implementation in an intervention trial. J Hum Nutr Diet. 2014 Oct;27(5):413-25. doi: 10.1111/jhn.12158. Epub 2013 Sep 20. PMID 24112099
- [Result] Sen A, Ren J, Ruffin MT, Turgeon DK, Brenner DE, Sidahmed E, Rapai ME, Cornellier ML, Djuric Z. Relationships between serum and colon concentrations of carotenoids and fatty acids in randomized dietary intervention trial. Cancer Prev Res (Phila). 2013 Jun;6(6):558-65. doi: 10.1158/1940-6207.CAPR-13-0019. Epub 2013 Apr 16. PMID 23592741
- [Result] Umoh FI, Kato I, Ren J, Wachowiak PL, Ruffin MT 4th, Turgeon DK, Sen A, Brenner DE, Djuric Z. Markers of systemic exposures to products of intestinal bacteria in a dietary intervention study. Eur J Nutr. 2016 Mar;55(2):793-798. doi: 10.1007/s00394-015-0900-7. Epub 2015 Apr 24. PMID 25903259
- [Result] Djuric Z, Turgeon DK, Ren J, Neilson A, Plegue M, Waters IG, Chan A, Askew LM, Ruffin MT 4th, Sen A, Brenner DE. Effects of a Mediterranean Diet Intervention on Anti- and Pro-Inflammatory Eicosanoids, Epithelial Proliferation, and Nuclear Morphology in Biopsies of Normal Colon Tissue. Nutr Cancer. 2015;67(5):721-9. doi: 10.1080/01635581.2015.1029637. Epub 2015 Apr 14. PMID 25869112
- [Result] Li Y, Sen A, Ren J, Askew LM, Sidahmed E, Brenner DE, Ruffin MT 4th, Turgeon DK, Djuric Z. Effects of vitamin E from supplements and diet on colonic alpha- and gamma-tocopherol concentrations in persons at increased colon cancer risk. Nutr Cancer. 2015;67(1):73-81. doi: 10.1080/01635581.2015.965333. Epub 2014 Nov 5. PMID 25372556
- [Result] Porenta SR, Ko YA, Gruber SB, Mukherjee B, Baylin A, Ren J, Djuric Z. Interaction of fatty acid genotype and diet on changes in colonic fatty acids in a Mediterranean diet intervention study. Cancer Prev Res (Phila). 2013 Nov;6(11):1212-21. doi: 10.1158/1940-6207.CAPR-13-0131. Epub 2013 Sep 10. PMID 24022589
- [Derived] Djuric Z, Bassis CM, Plegue MA, Ren J, Chan R, Sidahmed E, Turgeon DK, Ruffin MT 4th, Kato I, Sen A. Colonic Mucosal Bacteria Are Associated with Inter-Individual Variability in Serum Carotenoid Concentrations. J Acad Nutr Diet. 2018 Apr;118(4):606-616.e3. doi: 10.1016/j.jand.2017.09.013. Epub 2017 Dec 21. PMID 29274690
- [Derived] Sidahmed E, Sen A, Ren J, Patel A, Turgeon DK, Ruffin MT, Brenner DE, Djuric Z. Colonic Saturated Fatty Acid Concentrations and Expression of COX-1, but not Diet, Predict Prostaglandin E2 in Normal Human Colon Tissue. Nutr Cancer. 2016 Oct;68(7):1192-201. doi: 10.1080/01635581.2016.1213866. Epub 2016 Aug 22. PMID 27548026

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Healthy Eating: Healthy People 2010 Diet
  Healthy People 2010 Diet through dietary counseling: 6 months telephone counseling
- 2 Mediterranean: Mediterranean Diet
  Mediterranean Diet through dietary counseling: 6 months telephone counseling
Period: Overall Study
Arm/Group | 1 Healthy Eating | 2 Mediterranean
Started | 61 | 59
Completed | 46 | 47
Not Completed | 15 | 12
Not completed — Withdrawal by Subject | 12 | 12
Not completed — Protocol Violation | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Healthy Eating | 2 Mediterranean | Total
Number analyzed (Participants) | 61 | 59 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13) | 55 (10) | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 43 | 86
  Male | 18 | 16 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 61 | 58 | 119
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 55 | 52 | 107
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 59 | 120

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Dietary Goals
Description: Percentage of participants who met 70% of diet goals as outlined in the exchange list
Time Frame: 6 months
Measure: Number; unit: percentage of participants meeting goals
Arm/Group | 1 Healthy Eating | 2 Mediterranean
Number analyzed (Participants) | 61 | 59
percentage of participants meeting goals | 89 | 85

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | 1 Healthy Eating | 2 Mediterranean
Serious Adverse Events (participants affected / at risk) | 0/61 | 2/59
Other Adverse Events (participants affected / at risk) | 15/61 | 18/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Healthy Eating (N=61) | 2 Mediterranean (N=59)
surgery (Gastrointestinal disorders) | 0 (0) | 1 (1) — bowel obstruction
bipolar relapse (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Healthy Eating (N=61) | 2 Mediterranean (N=59)
various minor conditions (Infections and infestations) | 15 (15) | 18 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No